CLINICAL TRIAL: NCT07051291
Title: The Acute Effect of Instant Coffee in Different Forms on Plasma Metabolites
Brief Title: Acute Effects of Instant Coffee in Capsule vs Beverage Form on Plasma Metabolites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Seow Wei Jie, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NUS-IRB-2021-464
Record Dates: First submitted 2025-06-01; First posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Coffee

STUDY DESIGN:
Intervention Model Description: Participants will receive both interventions (instant coffee capsule and instant coffee beverage) in a randomized order across two visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Instant coffee capsule/ coffee beverage (Experimental)
  Interventions: Dietary Supplement: Instant Coffee Capsule; Dietary Supplement: Instant Coffee Beverage
- Instant coffee beverage/ coffee capsule (Experimental)
  Interventions: Dietary Supplement: Instant Coffee Capsule; Dietary Supplement: Instant Coffee Beverage

INTERVENTIONS:
Dietary Supplement: Instant Coffee Capsule — Participants received 1.7 grams of instant coffee in the form of three capsules. 200 mL of plain water was provided to participants to swallow the three capsules.
Dietary Supplement: Instant Coffee Beverage — Dissolved 1.7 grams of instant coffee in 200 mL of hot water to make a coffee beverage.

SUMMARY:
This study is designed to evaluate the acute effect of consuming a cup of instant coffee on circulating metabolites and to evaluate whether ingestion of instant coffee in the form of a capsule has a similar effect on circulating metabolites as compared to the conventionally prepared beverage.

ELIGIBILITY:
Inclusion Criteria: Healthy individuals aged 21-64 years old of Chinese ethnicity and are physically-abled, can participate in the research, and are able to understand English

Exclusion Criteria:

* Pregnant or breastfeeding
* Certain medications including Zanaflex, Sirasalud, Ketanest S, Spravato and Ephedrine Sulfate
* Any pre-existing medical conditions, depression, anxiety, caffeine/lactose intolerant, fear of needles and/or blood disorders, allergy to coffee or bovine capsules
* Existing dietary restrictions which makes them unable to consume non-halal certified bovine gelatin (the capsule encasing the coffee powder)
* Recent history of major surgical operations in the past year
* Past or current user of oral/systemic hormone treatment or therapies
* Taken antibiotics in the last 3 months
* Taking nutritional supplements (that contains coffee/tea-related compounds naturally found in other plants)
* Not willing to travel to the University for the study
* Unable to commit to completing both study visits

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2020-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Caffeine and polyphenol metabolites | The period between the two study visits ranged between 7 to 28 days.
  Each participant underwent two interventions, and blood was collected pre- and post- each intervention. Blood was allowed to clot at room temperature. After 30-40 min, serum was separated from entire blood by centrifugation (3000g, 15 min, 4°C) and aliquoted into tubes. All samples were processed on the same day of collection. A total of 7 biomarker compounds (trigonelline, paraxanthine, theophylline, theobromine, caffeine, cyclo(Leu-Pro), and cyclo(Pro-Val)) were quantified using a targeted method developed in-house. The quantification method was optimized by LC retention elution, parent-daughter quantifier mass transitions, and varying MS cone and collision energies (in V) to obtain clear peak separation and height. Multiple Reaction Monitoring (MRM) in positive electrospray ionization mode was performed on a Waters Xevo TQ-S Triple Quadrupole Mass Spectrometer system.

CONTACTS AND LOCATIONS:
Locations (1):
- Saw Swee Hock School of Public Health, National University of Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-23): https://cdn.clinicaltrials.gov/large-docs/91/NCT07051291/Prot_SAP_000.pdf